CLINICAL TRIAL: NCT06870721
Title: Long Head of Biceps as an Anterior Dynamic Sling for Recurrent Anterior Shoulder Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed hussein khalil, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-208-2024
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Dislocation
Keywords: Dynamic anterior stabilization; onlay; glenohumeral instability.
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: case series of 25 patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arthroscopic dynamic anterior stabilization for recurrent anterior shoulder dislocation (Experimental): arthroscopic dynamic anterior stabilization using Long head of biceps as for recurrent anterior shoulder dislocation arthroscopic transfer of the Long head of biceps to the anterior glenoid inpatients with recurrent shoulder dislocation
  Interventions: Procedure: arthroscopic dynamic anterior stabilization for recurrent anterior shoulder dislocation

INTERVENTIONS:
Procedure: arthroscopic dynamic anterior stabilization for recurrent anterior shoulder dislocation — arthroscopic dynamic anterior stabilization transferring long head of biceps to the anterior glenoid in patients with recurrent anterior shoulder dislocation

SUMMARY:
Purpose: To evaluate the functional outcomes of arthroscopic onlay dynamic anterior stabilization (DAS) using the long head of biceps (LHB) tendon for treatment of anterior glenohumeral instability (AGI) with limited to subcritical glenoid bone loss (GBL).

DETAILED DESCRIPTION:
Twenty-five patients underwent arthroscopic DAS using LHB between March 2022 and October 2022 for treatment of anterior glenohumeral instability (AGI) with limited to subcritical glenoid bone loss (GBL) were included in a prospective study with a minimum follow-up period of 2 years. The shoulder functional outcomes were assessed using the Rowe and the Quick Disabilities of Arm, Shoulder and Hand (Quick DASH) scores both preoperative and at 2 years follow-up. Magnetic resonance imaging (MRI) at 6 months after surgery to evaluate LHB tendon healing to the anterior glenoid.

ELIGIBILITY:
The inclusion criteria were

* Patients complaining of AGI, with one or more events of anterior shoulder dislocation.
* Associated limited (<13.5%) to subcritical (<25%) GBL.
* Positive anterior shoulder apprehension.

The exclusion criteria were

* Associated critical GBL (≥25%).
* Concomitant LHB lesion or rupture.
* Multidirectional or voluntary shoulder instability.
* Prior arthroscopic shoulder stabilization procedure.
* Concomitant rotator cuff tears.
* Acute proximal humerus fractures of the involved shoulder.

Ages: 20 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
rowe score | baseline, and 2 years postoperative
  shoulder score, the maximum is 100, the minimum is zero, the higher score means a better outcome
Quick Disabilities of Arm, Shoulder and Hand | baseline, and 2 years postoperative
  shoulder score, the maximum is 100, the minimum is zero, the higher score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H khalil, M.D, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu C, Xu J, Fang Z, Chen J, Ye Z, Wang L, Kang Y, Zhao S, Xu C, Zhao J. Arthroscopic Dynamic Anterior Stabilization Using Either Long Head of the Biceps or Conjoined Tendon Transfer for Anterior Shoulder Instability Results in a Similarly Low Recurrence Rate. Arthroscopy. 2023 Jul;39(7):1618-1627. doi: 10.1016/j.arthro.2022.12.040. Epub 2023 Jan 25. PMID 36708745
- [Background] Collin P, Nabergoj M, Denard PJ, Wang S, Bothorel H, Ladermann A. Arthroscopic Biceps Transfer to the Glenoid With Bankart Repair Grants Satisfactory 2-Year Results for Recurrent Anteroinferior Glenohumeral Instability in Subcritical Bone Loss. Arthroscopy. 2022 Jun;38(6):1766-1771. doi: 10.1016/j.arthro.2021.11.043. Epub 2021 Dec 7. PMID 34883198
- [Background] de Campos Azevedo C, Angelo AC. Onlay Dynamic Anterior Stabilization With Biceps Transfer for the Treatment of Anterior Glenohumeral Instability Produces Good Clinical Outcomes and Successful Healing at a Minimum 1 Year of Follow-Up. Arthrosc Sports Med Rehabil. 2023 Feb 23;5(2):e445-e457. doi: 10.1016/j.asmr.2023.01.012. eCollection 2023 Apr. PMID 37101880
- [Background] Milenin O, Toussaint B. Labral Repair Augmentation by Labroplasty and Simultaneous Trans-Subscapular Transposition of the Long Head of the Biceps. Arthrosc Tech. 2019 Apr 26;8(5):e507-e512. doi: 10.1016/j.eats.2019.01.010. eCollection 2019 May. PMID 31194141